CLINICAL TRIAL: NCT06030310
Title: Effects of the Application of a Motor Programme Throughout an Academic Year on the Neurological Maduration of a Sample of 2nd Grade Children of Primary Schools in Catalonia
Brief Title: Effects of Application of a Motor Programme on Neurological Maduration in Children
Acronym: Move&Learn
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Universitària del Bages (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: UManresa_Move&Learn 2023
Record Dates: First submitted 2023-07-25; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Child Development
Keywords: Primitive reflex; Motor function; Oculomotor function; Risk of presenting dyslexia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INPP Movement Program Group (Experimental): The INPP Movement Program Group will consist on a group of children aged between 7 and 9 years old enrolled in the second grade class of a catalan school that will participate in the school motor program provided by the Institute of Neuro-Physiology Psychology (INPP). This program consists of exercises that replicate the developmental movements of babies. Each day, a set of specific exercises will be performed, it will be practiced for 6 weeks and replaced by another set of exercises. They will be conducted for 15 minutes daily throughout the entire academic year.
  Interventions: Other: The developmental Exercise Programme of INPP
- Non Intervention Group (No Intervention): Children aged between 7 and 9 years old enrolled in the second grade at a catalan school. Students in the Non Intervention Group will continue with their regular academic school year without any additional intervention. If any student from the INPP Movement Program Group chooses not to participate in the study, they will join the class of the Non Intervention Group during the time when their peers are engaged in the school motor program.

INTERVENTIONS:
Other: The developmental Exercise Programme of INPP — The INPP school motor program consists of a series of developmental movements based on the normal movements of a child in their first year of life. Exercises must be performed as slow as possible and must be repeated for at least six weeks.
  Once the children have performed a set of movements, a new set will be presented for practice in a more complex position.
  The exercises are done on the floor and aid in developing:
  Proper alignment of the head with the body, trunk stability. Balance and coordination. The ability to use both sides of the body and upper and lower parts independently.
  Muscle tone in prone and supine position. Hand-eye coordination and visual skills
  Arms: INPP Movement Program Group

SUMMARY:
The persistence of primitive reflexes in school-age children can affect neuromotor maturation. Some studies link the persistence of primitive reflexes with specific learning difficulties, low academic performance, neurodevelopmental disorders, and behavioral problems. There are studies that suggest introducing intervention programs to help integrate the activity of these reflexes. The objective of this study is to assess the effects of implementing a motor program on the neurologic maturation of second-grade children throughout an academic year in Catalonia.

A prospective experimental longitudinal and randomized pre-post study will be conducted with two groups: Non Intervention group and intervention group, known as the INPP Movement Program Group (with daily application of the motor program), lasting for one academic year (from September '23 to June '24). Currently, a feasibility study will be conducted at a school in Valls, with a sample of 50 children, and data will be collected at the beginning and end of the academic year. The study will analyze primitive reflexes, motor skills related to balance and coordination, oculo-motor skills, and the risk of presenting dyslexia. Once the feasibility study is completed, the same study with appropriate modifications will be carried out in different schools across Catalonia during the academic year 2024 - 2025 (yet to be determined).

DETAILED DESCRIPTION:
Introduction: In a study conducted in Catalonia in 2020, it was found that 18,3% of school-age children between 5 and 17 years old had some neurodevelopmental disorder. There are studies that relate neurodevelopment to neuromotor immaturity and the presence of primitive reflexes. Others studies associate primitive reflexes with: attention deficit (ADD), attention deficit/hyperactivity disorder (ADHD), motor disorders and cognitive performance disorders.

Neuromotor immaturity, as defined by The Institute for Neuro-Physiological Psychology (INPP), involves the retention of a set of primitive reflexes beyond the first year of life and the absence and/or underdevelopment of postural reflexes beyond three years of age.

Primitive reflexes promote movement, and through movement, these reflexes gradually integrate. As a result, primitive reflexes are replaced by more mature postural reactions that are used throughout life. Properly developed postural reactions form the basis of good posture, balance, and coordination. However, in older age, some primitive reflexes may remain unintegrated. Regardless of a child's age, the presence of these reflexes indicates neuromotor immaturity.

Some studies describe primitive reflexes as one of the contributing factors to neurodevelopmental disorders, affecting the harmonious motor development of the child. Immature motor skills have been linked to learning difficulties such as reading and writing problems, difficulties in numerical skills, dyslexia, and behavioral problems. The presence of retained primitive reflexes is more common in children with neurodevelopmental disorders, and it acts as a barrier to learning.

There is evidence linking the presence of primitive reflexes to visual skills in children aged 6 to 14 years. Visual skills can influence reading and writing due to the connection between visual skills and hand-eye coordination. These visual skills, along with balance, coordination, and postural control, are essential for fixing the gaze and reading and writing fluently.

Studies have shown that by reducing the presence of primitive reflexes through motor activity, learning difficulties can also be reduced, leading to improved academic performance in students.

In 1996, INPP developed a school program intended to be applied collectively in classrooms with the aim of reducing neuromotor immaturity in students aged 7 and above. This school program designed by INPP consists of two parts: the INPP Test Battery for schools and the INPP motor exercise program. The INPP Test Battery for schools comprises a set of tests to evaluate the presence of unintegrated primitive reflexes and psychomotor skills (primarily related to aspects of balance and coordination). The INPP motor exercise program consists of a set of exercises designed to replicate the developmental movements of infants during early stages of neurodevelopment. This assessment and therapeutic tool can be used by various professionals, but it is specifically designed for teachers and other professionals involved in education and child development to identify and treat children displaying signs of neuromotor immaturity. This tool has not been validated in English, Spanish, or Catalan.

Some studies have applied motor programs to reduce the presence of primitive reflexes and have shown improvements in the maturation of primitive reflexes. These programs are proposed as possible ways to address neuromotor immaturity.

There is limited evidence on the relationship between motor function, primitive reflexes, and learning impairments. A review on these three aspects, published in 2022, recommends further research on the topic.

Hypothesis: Implementing the INPP school program in classrooms for second-grade students in Catalan schools will enable the assessment and integration of remaining primitive reflexes, leading to improvements in neuro-motor maturation, oculomotor skills, and a reduction in the incidence of risk of dyslexia.

Objectives: After completing Phase 1, which involved a viability test of selected evaluation tools (April 2023), the objective is to initiate Phase 2:

Phase 2: Prospective experimental longitudinal non-randomized study with two groups: Non Intervention group and intervention group, known as the INPP Movement Program Group (with daily application of the motor program). The study will be conducted in second-grade students at Claret School in Valls. Both groups will undergo the INPP school program assessment battery and specific tests to evaluate oculomotor skills and the risk of dyslexia at the beginning and end of the school year. The INPP Movement Program Group will perform the INPP motor program for 15 minutes daily throughout the academic year, while the Non Intervention Group will continue their regular school curriculum without the specific motor program but may receive it in the following academic year (2024-25) if significant benefits for students are demonstrated.

This school program only excludes those children who have difficulties in performing the exercises (e.g., due to a motor impairment) or those who cannot understand the instructions and thus cannot be evaluated with the pre-program motor assessments (e.g., newcomers who don't understand the language).

Phase 3: Prospective experimental longitudinal study in different schools in Catalonia, each with a significant sample size, to assess neuromotor maturation pre- and post-application of the INPP school program in relation to different variables: primitive reflexes, oculomotor skills, and the risk of dyslexia in children.

Ethical Aspects:

This project has undergone evaluation by an ethics committee, and a favorable opinion was obtained in November 2022.

The legal guardians of the study participants will be informed through an information sheet prior to their inclusion and through an informative meeting that will take place at the schools. These guardians will sign the informed consent sheet. As this study involves child participants, the informed consent will be signed by the legal guardian.

Due to the nature of the study and its methodological phases, it is not anticipated that there will be any health risks to the participants during its execution. Moreover, those who wish to do so can withdraw from the study at any time without any negative repercussions.

At the end of the study, schools and/or families that wish to do so will receive a summary of the obtained results and publications resulting from the study, upon request to the principal investigator.

In the next school year, the option of applying the school program will be offered to the control group that did not receive it during the study.

All data will be coded, meaning each participant will be assigned a code, and it will be impossible to identify participants with the given responses, ensuring confidentiality. At all times, the General Data Protection Regulation (EU) 2016/679, the Data Protection Act (GDPR), Organic Law 3/2018, December 5, on personal data protection and guarantee of digital rights, and Organic Law 1/1982, May 5, on the protection of the civil right to honor, personal and family privacy, and one's own image will be respected. Additionally, the guidelines of the Code of Ethics of the College of Physiotherapists and the Declaration of Helsinki on human rights in medical research will be followed.

The data will be stored by the principal investigator in the OneDrive of the Fundació Universitària del Bages Campus Manresa of the UVic-UCC, linked to the project. The coded database will only be accessible to the research team members who need to analyze the results through a personalized and temporary link to the OneDrive of the Fundació Universitària del Bages Campus Manresa of the Uvic-UCC or on the laptop safeguarded by the principal investigator.

No recordings will be made as they are not essential for the study.

ELIGIBILITY:
Inclusion Criteria:

* Children enrolled in the second grade of the selected schools
* Age between 7 and 9 years

Exclusion Criteria:

* Children unable to perform the exercises due to physical and/or cognitive limitations
* Those unable to consistently attend the therapy sessions (with an absence rate of more than 80%) or have physical limitations
* Children who cannot understand the language and therefore cannot complete the questionnaires and tests to be conducted

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2023-06-10 (Actual); Primary Completion 2024-06-20 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Reflex status | At the begining and at the end of an academic year
  To assess the neuromotor maturation pre and post application of the INPP school programme in 2nd grade children of different schools in Catalonia and its relation to reflex status using the INPP Test battery for use in schools.
  The Test battery consists on:
  Ayres Test for the Asymmetric Tonic Neck Reflex Hoff -Schilder Test for the The Asymmetric Tonic Neck Reflex Ayres Test for the Symmetric Tonic Neck Reflex Erect Test for the Tonic Labyrinth Reflex
  The assessment is through a 5-point likert scale where 0 means no retention of primitive reflexes and no immaturity and 5 means 100% dysfunction.

SECONDARY OUTCOMES:
Motor skills | At the begining and at the end of an academic year
  To assess the neuromotor maturation pre and post application of the INPP school programme in 2nd grade children of different schools in Catalonia and its relation to motor skills
  To assess the motor skills it will be used the Movement Battery Assesment for children (MABC Test) internationally used to detect developmental coordination disorders (DCD)
  The test has three specific dimensions of the child motor skills:
  Hand dexterity Catching and aiming Balance. The assessment is through a 5-point likert scale where 0 means no disfunction and and 5 means 100% dysfunction.
oculomotor functioning | At the begining and at the end of an academic year
  To assess the neuromotor maturation pre and post application of the INPP school programme in 2nd grade children of different schools in Catalonia and its relation to oculomotor functioning
  To assess the oculomotor functioning it will be used the Developmental Eye Movement Test (DEM).
  It´s a battery that includes three subtests to assess vertical and horizontal eye movements.
  The evaluation is through 3 variables to be calculated for each child: horizontal time, vertical time and the ratio between both.
  These results related to a range of age are compared with the table of the average values (table from 7 to 7 years and 11 months with its categorisation).
risk of presenting dyslexia. | At the begining and at the end of an academic year
  To assess the neuromotor maturation pre and post application of the INPP school programme in 2nd grade children of different schools in Catalonia and its relation to the measure of risk of presenting dyslexia.
  The tool to assess the risk of dyslexia is the Spanish Test Battery called Diagnosis and Early Detection of Dyslexia (PROLEXIA) designed to cover two main purposes: early detection and differential diagnostic testing to assess the risk of dyslexia.
  The categorisation of prolexia risk ranges from very low risk (0 points) to very high risk (more than 200 points), through low ( 35-55), moderate ( 55-75) and high ( 75-110).

CONTACTS AND LOCATIONS:
Overall Officials: Marta Not Monegal, MSc, Principal Investigator — University of Vic - Central University of Catalonia
Locations (1):
- Marta Not Monegal, Manresa, Barcelona, Spain

REFERENCES:
- [Background] McWhirter K, Steel A, Adams J. The association between learning disorders, motor function, and primitive reflexes in pre-school children: A systematic review. J Child Health Care. 2024 Jun;28(2):402-428. doi: 10.1177/13674935221114187. Epub 2022 Jul 13. PMID 35830652
- [Background] Pecuch A, Gieysztor E, Wolanska E, Telenga M, Paprocka-Borowicz M. Primitive Reflex Activity in Relation to Motor Skills in Healthy Preschool Children. Brain Sci. 2021 Jul 23;11(8):967. doi: 10.3390/brainsci11080967. PMID 34439585
- [Background] Gieysztor EZ, Choinska AM, Paprocka-Borowicz M. Persistence of primitive reflexes and associated motor problems in healthy preschool children. Arch Med Sci. 2018 Jan;14(1):167-173. doi: 10.5114/aoms.2016.60503. Epub 2016 Jun 13. PMID 29379547
- See also: The association between learning disorders, motor function, and primitive reflexes in pre-school children: A systematic review. — https://pubmed.ncbi.nlm.nih.gov/35830652/
- See also: Primitive Reflex Activity in Relation to Motor Skills in Healthy Preschool Children — https://pubmed.ncbi.nlm.nih.gov/34439585/
- See also: Persistence of primitive reflexes and associated motor problems in healthy preschool children. — https://pubmed.ncbi.nlm.nih.gov/29379547/